CLINICAL TRIAL: NCT06636838
Title: Language Matters: Exploring the Impact of Language Concordance on Fertility Treatment Progression
Acronym: ImpaLa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB ID #: 202407176
Record Dates: First submitted 2024-09-30; First posted 2024-10-15 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Infertility; Infertility (IVF Patients); Infertility Assisted Reproductive Technology; Ovulation Ind
Keywords: Spanish speaking; Spanish; infertility; Infertility work-up; IVF
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spanish speaking patients seen by English-Speaking Provider (No Intervention): Spanish speaking patients will be seen by our English-speaking providers using a qualified interpreter.
- Spanish-Speaking patients seen by a Spanish-speaking provider (Experimental): Spanish speaking patients will be seen by our Spanish-speaking provider
  Interventions: Behavioral: Spanish-Speaking Provider

INTERVENTIONS:
Behavioral: Spanish-Speaking Provider — Spanish speaking patients will be seen by our Spanish-speaking provider
  Arms: Spanish-Speaking patients seen by a Spanish-speaking provider

SUMMARY:
Currently, patients presenting to the Fertility and Reproductive Medicine Center meet with an English-speaking provider and communicate through an interpreter, as none of the physicians speak Spanish. However, this study PI is a native Spanish speaker and certified bilingual clinician. Thus, this study is looking to evaluate whether or not the use of an interpreter delays completion of testing and initiation of fertility treatment. The medically indicated testing, procedures, and course of treatment will not be altered as a result of participation in the study. Participants will be asked to complete a survey in their preferred language to gauge satisfaction and communication efficacy.

This proposed study is significant as it seeks to address a critical gap in the understanding of how language concordance between healthcare providers and patients influences treatment outcomes in fertility care. With Spanish being the most commonly spoken non-English language in the U.S., evaluating the impact of Spanish language skills in medical care is both timely and essential. This research will shed light on whether Spanish-speaking patients experience better treatment progression and outcomes when cared for by language-concordant providers versus when interpreters are used in fertility care.

This prospective study will be conducted at Washington University's Fertility and Reproductive Medicine Center over a 12-month period. The investigators aim to enroll a total of 70 Spanish-speaking patients, based on previous patient trends at the Center 35 will be randomized to the intervention group (being evaluated and treated by a Spanish-speaking provider), and 35 will be randomized to standard of care (communicating with an English-speaking provider through an interpreter).

ELIGIBILITY:
Inclusion Criteria:

* Must be greater than 18 years old
* Preferred language must be Spanish speaking
* Must be seeking fertility treatment

Exclusion Criteria:

* Preferred language English
* Not currently seeking fertility care
* Less than 18 years old

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Completion of diagnostic tests | 90 days from initial consultation.
  The primary outcome is the time from the patients initial consultation to the completion of the recommended fertility diagnostic tests such as blood work or a pelvic ultrasound. Given that the tests are typically specific to the menstrual cycle, the investigators want know if the patients are completing their work-up faster when they see a Spanish-speaking physician thus understanding the instructions versus when the English speaking providers use an interpreter. The work-up only includes the labs and imaging that was recommended during their initial visit. The outcome will be measured by the unit - days.

SECONDARY OUTCOMES:
Patient satisfaction and communication | 90 days from initial consultation.
  Patient satisfaction and communication effectiveness, assessed through surveys administered after the initial consultation. The survey is a validated survey that uses a point system metric to conclude patient satisfaction similar to the PHQ-9 survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jain M, Peterson A, Nguyen N, Goldsammler M. Reproductive inequity and inferior intrauterine insemination outcomes in patients with limited English proficiency: a retrospective cohort study. Fertil Steril. 2023 Oct;120(4):844-849. doi: 10.1016/j.fertnstert.2023.05.154. Epub 2023 May 22. PMID 37225071
- [Background] Lopez Vera A, Thomas K, Trinh C, Nausheen F. A Case Study of the Impact of Language Concordance on Patient Care, Satisfaction, and Comfort with Sharing Sensitive Information During Medical Care. J Immigr Minor Health. 2023 Dec;25(6):1261-1269. doi: 10.1007/s10903-023-01463-8. Epub 2023 Feb 25. PMID 36840903
- [Background] Berdahl TA, Kirby JB. Patient-Provider Communication Disparities by Limited English Proficiency (LEP): Trends from the US Medical Expenditure Panel Survey, 2006-2015. J Gen Intern Med. 2019 Aug;34(8):1434-1440. doi: 10.1007/s11606-018-4757-3. Epub 2018 Dec 3. PMID 30511285
- See also: Language Use in the United States: 2019 — https://www.census.gov/content/dam/Census/library/publications/2022/acs/acs-50.pdf